CLINICAL TRIAL: NCT06687278
Title: The Effect of Interpersonal Relationship Psychotherapy-Based Intervention Program on Psychosocial Well-Being of Female Victims of Intimate Partner Violence
Brief Title: Effectiveness of Interpersonal Relationship Psychotherapy Intervention for Female Victims of Intimate Partner Violence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cennet Kara Özçalık, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUC-CKOzcalik-001
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Intimate Partner Violence (IPV); Interpersonal Psychotherapy; Interpersonal Relations
Keywords: Intimate Partner Violence; Psychological Well-Being; Interpersonal Relations; Interpersonal Psychotherapy; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will employ a pretest-posttest-follow-up test experimental design with a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Initiative Group (Experimental): Participants in this group will receive an Interpersonal Relationship Psychotherapy-Based Intervention Program consisting of eight individual sessions.
  Interventions: Behavioral: Interpersonal Relationship Psychotherapy-Based Intervention Program
- The Control Group (No Intervention): The control group will be left unaltered throughout the course of the study. In the event that participants are already undergoing medical and/or supportive care outside of the parameters of the study, they shall continue to receive such care according to standard protocols.

INTERVENTIONS:
Behavioral: Interpersonal Relationship Psychotherapy-Based Intervention Program — The Interpersonal Relationship Psychotherapy-Based Intervention Program is based on IPR and developed with reference to relevant literature and a previously published study (Cort et all., 2014). Subsequent to the development of the program, a series of expert opinions were obtained from seven specialists in the field. The Interpersonal Relationship Psychotherapy-Based Intervention Program is a 2.5-3 month program comprising eight individual sessions. The program is designed to be administered on a weekly basis, with each session lasting approximately 45-60 minutes. The participants in this group will receive an Interpersonal Relationship Psychotherapy Based Intervention Programme, which consists of eight individual sessions.
  Arms: The Initiative Group

SUMMARY:
This interventional study aims to examine the impact of the Interpersonal Relationship Psychotherapy-Based Intervention Program on the psychosocial well-being of female victims of intimate partner violence.

The main questions to be answered are the following:

1. Is the Interpersonal Relationship Psychotherapy-Based Intervention Program effective on the interpersonal problems of female victims of intimate partner violence?
2. Is the Interpersonal Relationship Psychotherapy-Based Intervention Program effective on the mental well-being of female victims of intimate partner violence?

The study will include eight individual interviews using a variety of data collection forms.

DETAILED DESCRIPTION:
World Health Organization, defines intimate partner violence as behaviours that cause physical, sexual or psychological harm in an intimate relationship. These behaviours include physical aggression, sexual coercion, psychological abuse and controlling behaviours. One in three women will experience violence from a partner at some point in their lifetime. A strong correlation has been identified between women's exposure to violence and their susceptibility to mental health issues. In instances of prolonged violence, women tend to exhibit a range of emotional responses, including feelings of insecurity, loss of control, guilt, low self-esteem, helplessness, and hopelessness.

Interpersonal Psychotherapy (IPT) is a time-limited psychotherapy developed in the 1970s for the treatment of depression. It focuses on interpersonal relationships and social support systems. The primary focus of IPT is on the resolution of existing interpersonal conflicts. IPT is delivered to different clinical populations across the lifespan in a range of flexible formats, including individual, couple, group, telephone sessions, and web-based applications in a variety of settings and doses. It has been demonstrated to be an efficacious intervention for the treatment of psychiatric disorders, including anxiety disorders, depression, post-traumatic stress disorder, and bipolar disorder, particularly during the perinatal period. Despite the existence of numerous studies examining the impact of IPT across diverse populations, only one investigation has explored the efficacy of IPT in women who have experienced violence. In the aforementioned examination, no established treatment program for women victims of intimate partner violence has been identified in our country. Although intimate partner violence affects a significant proportion of the population, the paucity of studies focusing on interpersonal relationships in this context represents a gap in the existing literature.

Given the high prevalence of violence against women and the associated burden of physical, mental, social, and social problems, as well as the limitations of existing intervention programs designed to enhance the psychosocial well-being of women victims of intimate partner violence, it is imperative to develop novel intervention strategies that prioritize interpersonal relationships and aim to bolster the coping skills and social support systems of these individuals. In light of the aforementioned considerations, the objective of the present study is to examine the impact of an intervention program based on interpersonal relationship psychotherapy on the psychosocial well-being of women victims of intimate partner violence. This study will examine the psychosocial well-being, interpersonal problems and mental well-being levels of women victims of intimate partner violence.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in the Turkish language, including the ability to speak and understand it.
* Exposure to any form of violence perpetrated by an intimate partner.

Exclusion Criteria:

* Exposure to violence by an individual other than an intimate partner for the purpose of maintaining group homogeneity.
* Presence of sensory loss, including but not limited to hearing and vision.
* Physical injury and/or disability resulting from violence that precludes participation in the intervention program.
* Diagnosis of schizophrenia spectrum disorders and other psychotic disorders.
* Presence of active self-destructive thoughts and/or plans.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The research is focused on adult female participants who have experienced violence perpetrated by an intimate partner. Consequently, only individuals of the female gender are eligible to participate.
Enrollment: 40 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Inventory of Interpersonal Problems Circumplex Scales (IIP-C) | The scale will be administered during the second individual interview of the intervention phase.
  The scale was developed by Alden and colleagues for the purpose of assessing interpersonal functioning in the context of personal stress and difficulties. The scale employs a 5-point Likert-type response format, comprising a total of 32 items that assess various domains of interpersonal functioning. The scale comprises eight subscales, each comprising four items. Higher scores on the total scale and its constituent subscales indicate elevated levels of interpersonal stress and the presence of specific interpersonal difficulties. The Turkish validity and reliability study was conducted by Akyunus and Gencoz (2016), and the total scale Cronbach's alpha coefficient was found to be 0.86. The scale has been demonstrated to possess sufficient validity and reliability to be employed in research on interpersonal attitudes and behaviours in Turkey and in clinical applications.
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | The scale will be administered during the second individual interview of the intervention phase.
  The scale was developed by Tennant and colleagues as a means of measuring the mental well-being levels of individuals. The scale employs a 5-point Likert scale, with a minimum score of 14 and a maximum score of 70. The scale is scored according to the following key: 1=strongly disagree, 2=disagree, 3=somewhat agree, 4=agree, 5=strongly agree. The scale comprises 14 items, with higher scores indicative of elevated levels of psychological well-being. The reliability of the scale was evaluated in studies conducted with individuals aged 16 and above. The Cronbach alpha coefficient for the scale was found to be 0.89. The test-retest reliability coefficient of the scale was found to be 0.83. The Turkish reliability and validity study of the scale was conducted by Keldal (2015). The Cronbach's Alpha internal consistency reliability coefficient of the Turkish version of the scale was found to be 0.92.
Inventory of Interpersonal Problems Circumplex Scales (IIP-C) | The scale will be administered at the close of the eighth session.
  The scale was developed by Alden and colleagues for the purpose of assessing interpersonal functioning in the context of personal stress and difficulties. The scale employs a 5-point Likert-type response format, comprising a total of 32 items that assess various domains of interpersonal functioning. The scale comprises eight subscales, each comprising four items. Higher scores on the total scale and its constituent subscales indicate elevated levels of interpersonal stress and the presence of specific interpersonal difficulties. The Turkish validity and reliability study was conducted by Akyunus and Gencoz (2016), and the total scale Cronbach's alpha coefficient was found to be 0.86. The scale has been demonstrated to possess sufficient validity and reliability to be employed in research on interpersonal attitudes and behaviours in Turkey and in clinical applications.
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | The scale will be administered at the close of the eighth session.
  The scale was developed by Tennant and colleagues as a means of measuring the mental well-being levels of individuals. The scale employs a 5-point Likert scale, with a minimum score of 14 and a maximum score of 70. The scale is scored according to the following key: 1=strongly disagree, 2=disagree, 3=somewhat agree, 4=agree, 5=strongly agree. The scale comprises 14 items, with higher scores indicative of elevated levels of psychological well-being. The reliability of the scale was evaluated in studies conducted with individuals aged 16 and above. The Cronbach alpha coefficient for the scale was found to be 0.89. The test-retest reliability coefficient of the scale was found to be 0.83. The Turkish reliability and validity study of the scale was conducted by Keldal (2015). The Cronbach's Alpha internal consistency reliability coefficient of the Turkish version of the scale was found to be 0.92.
Inventory of Interpersonal Problems Circumplex Scales (IIP-C) | The scale will be administered within the fourth week following the eighth session.
  The scale was developed by Alden and colleagues for the purpose of assessing interpersonal functioning in the context of personal stress and difficulties. The scale employs a 5-point Likert-type response format, comprising a total of 32 items that assess various domains of interpersonal functioning. The scale comprises eight subscales, each comprising four items. Higher scores on the total scale and its constituent subscales indicate elevated levels of interpersonal stress and the presence of specific interpersonal difficulties. The Turkish validity and reliability study was conducted by Akyunus and Gencoz (2016), and the total scale Cronbach's alpha coefficient was found to be 0.86. The scale has been demonstrated to possess sufficient validity and reliability to be employed in research on interpersonal attitudes and behaviours in Turkey and in clinical applications.
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | The scale will be administered within the fourth week following the eighth session.
  The scale was developed by Tennant and colleagues as a means of measuring the mental well-being levels of individuals. The scale employs a 5-point Likert scale, with a minimum score of 14 and a maximum score of 70. The scale is scored according to the following key: 1=strongly disagree, 2=disagree, 3=somewhat agree, 4=agree, 5=strongly agree. The scale comprises 14 items, with higher scores indicative of elevated levels of psychological well-being. The reliability of the scale was evaluated in studies conducted with individuals aged 16 and above. The Cronbach alpha coefficient for the scale was found to be 0.89. The test-retest reliability coefficient of the scale was found to be 0.83. The Turkish reliability and validity study of the scale was conducted by Keldal (2015). The Cronbach's Alpha internal consistency reliability coefficient of the Turkish version of the scale was found to be 0.92.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | in the second interview with the participant
  It is a self-report scale designed to assess vegetative, emotional, cognitive, and motivational symptoms of depression. The scale items are presented on a 4-point Likert scale, with responses ranging from "not at all" to "very much" (0-3). The scale comprises 21 items, and it has been suggested that a score of 17 or above may be indicative of above-normal depression. A study of the validity and reliability of the scale in a Turkish cultural context was conducted by Hisli (1989) with a sample of university students. The original version of the scale exhibited a Cronbach's alpha coefficient of 0.92, while the Turkish version demonstrated a coefficient of 0.80.
Beck Depression Inventory (BDI) | end of session 8
  It is a self-report scale designed to assess vegetative, emotional, cognitive, and motivational symptoms of depression. The scale items are presented on a 4-point Likert scale, with responses ranging from "not at all" to "very much" (0-3). The scale comprises 21 items, and it has been suggested that a score of 17 or above may be indicative of above-normal depression. A study of the validity and reliability of the scale in a Turkish cultural context was conducted by Hisli (1989) with a sample of university students. The original version of the scale exhibited a Cronbach's alpha coefficient of 0.92, while the Turkish version demonstrated a coefficient of 0.80.
Intervention Program Evaluation Form | end of session 8
  In order to evaluate the effectiveness of the intervention program, the researcher employed a 5-point Likert-type scale (1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, 5 = strongly agree), based on self-report and aligned with the content of the intervention program. It is intended that each participant in the intervention group will complete the form at the post-test and follow-up test.
Beck Depression Inventory (BDI) | The scale will be administered within the fourth week following the eighth session.
  It is a self-report scale designed to assess vegetative, emotional, cognitive, and motivational symptoms of depression. The scale items are presented on a 4-point Likert scale, with responses ranging from "not at all" to "very much" (0-3). The scale comprises 21 items, and it has been suggested that a score of 17 or above may be indicative of above-normal depression. A study of the validity and reliability of the scale in a Turkish cultural context was conducted by Hisli (1989) with a sample of university students. The original version of the scale exhibited a Cronbach's alpha coefficient of 0.92, while the Turkish version demonstrated a coefficient of 0.80.
Intervention Program Evaluation Form | The scale will be administered within the fourth week following the eighth session.
  In order to evaluate the effectiveness of the intervention program, the researcher employed a 5-point Likert-type scale (1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, 5 = strongly agree), based on self-report and aligned with the content of the intervention program. It is intended that each participant in the intervention group will complete the form at the post-test and follow-up test.

CONTACTS AND LOCATIONS:
Overall Officials: Cennet Kara Özçalık, Principal Investigator — Istanbul Universty-Cerrahpasa
Locations (1):
- Florence Nightingale Faculty of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The requisite legal and ethical permissions for the research were obtained on the condition that the data would not be shared with third parties.

REFERENCES:
- [Background] Ruiz-Perez I, Plazaola-Castano J. Intimate partner violence and mental health consequences in women attending family practice in Spain. Psychosom Med. 2005 Sep-Oct;67(5):791-7. doi: 10.1097/01.psy.0000181269.11979.cd. PMID 16204440
- [Background] Mufson, L., Dorta, K.P., Moreau, D. and Weissman, M.M., 2004, Interpersonal Psychotherapy for Depressed Adolescents, 2nd ed., The Guilford Press, New York, ISBN-13: 978-1-59385-042-5.
- [Background] Ravitz P, Watson P, Lawson A, Constantino MJ, Bernecker S, Park J, Swartz HA. Interpersonal Psychotherapy: A Scoping Review and Historical Perspective (1974-2017). Harv Rev Psychiatry. 2019 May/Jun;27(3):165-180. doi: 10.1097/HRP.0000000000000219. PMID 30883446
- [Background] Cort, N. A., Cerulli, C., Poleshuck, E. L., Bellenger, K. M., Xia, Y., Tu, X., Mazzotta, C. M. and Talbot, N. L., 2014, Interpersonal psychotherapy for depressed women with histories of intimate partner violence, Psychological trauma: theory, research, practice, and policy, 6 (6), 700-707.
- [Background] Almis BH, Kutuk EK, Gumustas F, Celik M. Risk Factors for Domestic Violence in Women and Predictors of Development of Mental Disorders in These Women. Noro Psikiyatr Ars. 2018 Mar 19;55(1):67-72. doi: 10.29399/npa.19355. eCollection 2018 Mar. PMID 30042644
- [Background] Almis BH, Gumustas F, Kutuk EK, 2020, Effects of Domestic Violence Against Women on Mental Health of Women and Children, Current Approaches in Psychiatry, 12 (2), 232-242. doi: 10.18863/pgy.567635
- [Background] Atar, A.O. & Aydın, P.C., 2019, Evidence for Efficacy of interpersonal psychotherapy, Interpersonal Relations Psychotherapy, In Aydın, N., Omay, O. (ed), Türkiye Clinics, Ankara, 1st ed., 12-18.
- [Background] Akyunus, M., & Gencoz, T., 2016, Psychometric properties of the Inventory of Interpersonal Problems Circumplex Scales short form: a reliability and validity study, Dusunen Adam The Journal of Psychiatry and Neurological Sciences, 29 (1), 36-48. DOI: 10.5350/DAJPN2016290104
- [Background] Alden LE, Wiggins JS, Pincus AL. Construction of circumplex scales for the Inventory of Interpersonal Problems. J Pers Assess. 1990 Winter;55(3-4):521-36. doi: 10.1080/00223891.1990.9674088. No abstract available. PMID 2280321
- [Background] Keldal, G., 2015, Turkish Version of the Warwick-Edinburgh Mental Well-Being Scale: A validity and reliability study, The Journal of Happiness & Well-Being, 3 (1), 103-115.
- [Background] Hisli, N., 1989, Validity and reliability of Beck Depression Inventory for university students, Journal of Psychology, 7 (23), 3-13.
- [Background] Turgut EO, Cam MO. The Effect of Tidal Model-Based Psychiatric Nursing Approach on the Resilience of Women Survivors of Violence. Issues Ment Health Nurs. 2020 May;41(5):429-437. doi: 10.1080/01612840.2019.1672222. Epub 2020 Mar 18. PMID 32186926
- See also: World Health Organization (WHO), 2022, Intimate Partner Violence — https://apps.who.int/violence-info/intimate-partner-violence/
- See also: UN Women, 2021, Justice for women: High-level Group report — https://www.unwomen.org/en/digital-library/publications/2020/03/justice-for-women-high-level-group-report